CLINICAL TRIAL: NCT06958380
Title: The Impact of Corrective Exercise and Rehabilitation on a Patient With Fanconi Anemia: A Clinical Case Study
Brief Title: Corrective Exercise and Rehabilitation in Fanconi Anemia: A Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PA25FA-2-03
Record Dates: First submitted 2025-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Fanconi Anemia
Keywords: Corrective Exercise; Quality of Life (QoL); Physical Therapy Intervention; Fatigue; Postural Correction
MeSH Terms: conditions — Fanconi Anemia; Fatigue | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This is a longitudinal single-subject case study in which one adult patient diagnosed with Fanconi anemia will undergo a structured, in-person supervised corrective exercise and rehabilitation program. The subject will serve as their own control, with baseline measurements compared to post-intervention outcomes.
Masking Description: Due to the nature of a single-case study and individualized delivery of the intervention, blinding is not applicable. However, efforts will be made to minimize bias during outcome evaluation by having outcome measures reviewed by an independent assessor when possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): The patient in this clinical case study will undergo a 12-week corrective exercise and rehabilitation program specifically tailored to individuals with Fanconi Anemia. Each session will be conducted via in-person supervised sessions and will last approximately 40-45 minutes, performed three times per week, totaling 36 sessions. The program will incorporate exercises targeting postural correction, functional mobility, strength, and endurance, and will be supervised in real-time by a trained rehabilitation specialist.
  Interventions: Behavioral: Corrective exercise and rehabilitation

INTERVENTIONS:
Behavioral: Corrective exercise and rehabilitation — This is a longitudinal single-subject case study in which one adult patient diagnosed with Fanconi anemia will undergo a structured, supervised corrective exercise and rehabilitation program. The subject will serve as their own control, with baseline measurements compared to post-intervention outcomes.

SUMMARY:
Introduction: Fanconi anemia (FA) is a rare autosomal recessive DNA repair disorder characterized by congenital malformations, progressive bone marrow failure, and reduced quality of life. Although physical and occupational therapy are routinely recommended to address skeletal anomalies in FA, no studies have evaluated the impact of a structured corrective exercise and rehabilitation program on patient outcomes.

Method: In this single case clinical report, an adult FA patient will complete a 12 week supervised corrective exercise and rehabilitation program (36 sessions; 3 × 40-45 min/week) delivered via in-person supervised sessions. Primary outcome is change in patient reported quality of life (SF 36) from baseline to week 12; secondary outcomes include muscle strength, fatigue severity, postural parameters, and hematological indices.

DETAILED DESCRIPTION:
Fanconi anemia (FA), first described in 1927 by Dr. Guido Fanconi, is a rare, inherited, autosomal recessive disorder affecting proteins involved in DNA repair and cell cycle regulation. This syndrome is characterized by congenital malformations (involving the limbs, skeletal system, kidneys and urinary structures, sensory organs (eyes and ears) and central nervous system), progressive bone marrow failure (aplastic anemia), increased cancer incidence (particularly head/neck epithelial cancers and acute myeloid leukemia (AML)) and a range of physical anomalies (including microcephaly and short stature).

Higher prevalence rates of FA have been observed in populations with a high incidence of consanguineous marriages, including South African Blacks, Turks, Saudi Arabians, Ashkenazi Jews and Iranians. Globally, the disorder affects approximately 1 in every 160,000 to 360,000 individuals, while the estimated carrier frequency is around 0.3%.

FA results from mutations in at least 22 genes involved in genomic stability and DNA repair. The majority of FA-related changes-accounting for more than 80%-are found in the FANCA, FANCG, and FANCC genes, whereas alterations in the remaining genes are comparatively rare.

The diagnosis of FA, though challenging due to variable expressiveness, relies on clinical suspicion confirmed through genetic analysis. FA should be suspected in cases of de novo bone marrow failure, especially in younger patients, or in the presence of spontaneous chromosomal breaks and certain cytogenetic abnormalities. Early diagnosis, while not currently improving cure rates, enables healthcare professionals to implement systematic follow-up protocols and timely interventions.

Therapeutic management of FA relies on vigilant, risk adapted monitoring of hematologic status-complete blood counts and bone marrow assessments are scheduled from every six months to six weeks based on cytopenia severity-to detect dysplasia or clonal abnormalities. Supportive care with red cell and platelet transfusions, infection prophylaxis, and occasional androgen therapy helps maintain blood counts while preparing for hematopoietic stem cell transplantation (HSCT). Transplantation, preferably before transfusion dependence or emergence of poor risk cytogenetic changes, offers the only curative approach to marrow failure. Simultaneously, long term surveillance addresses FA's systemic complications through regular cancer screenings and organ specific evaluations.

Despite the established role of physical and occupational therapy in managing skeletal abnormalities in FA, there is a notable scarcity of research specifically examining the effectiveness of structured exercise rehabilitation programs for this population. In a similar study, Ye et al. (2024) found that a structured exercise rehabilitation program improved quality of life, reduced fatigue, and enhanced physical performance in aplastic anemia patients undergoing HSCT. These promising outcomes support the potential benefit of a similar approach in Fanconi anemia patients. Based on the identified research gaps, the investigators hypothesize that a structured program of corrective exercise, physical therapy interventions, and rehabilitation will improve quality of life, physical function, and potentially influence hematological parameters in patients with Fanconi anemia.

The primary objective of this case study is to evaluate the effectiveness of these interventions on patient-reported quality of life. Secondary objectives include assessing improvements in muscle strength, fatigue levels, functional independence in activities of daily living, and monitoring potential changes in hematological indicators. Our intervention will encompass a structured exercise rehabilitation program beginning at an appropriate phase of treatment and continuing through a defined follow-up period. This case study aims to provide preliminary evidence to guide the development of comprehensive rehabilitation protocols specifically designed for the FA population, addressing both the skeletal abnormalities and the systemic manifestations of the condition.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Fanconi Anemia through genetic testing
* Age 18 years or older
* Medically stable and cleared for exercise participation by their physician
* Ability to provide informed consent
* Access to a smartphone, tablet, or computer with stable internet connection
* Willingness to participate in scheduled rehabilitation sessions over 12 weeks

Exclusion Criteria:

* Presence of unstable medical conditions (e.g., uncontrolled infections, recent surgery, severe cardiopulmonary issues)
* Cognitive impairments that interfere with understanding or performing exercise instructions
* Recent hematopoietic stem cell transplantation (within past 3 months)
* Concurrent participation in another structured physical rehabilitation program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2025-05-03 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of changes in hyper-kyphosis | Pre-intervention and Week 12
  Evaluating the effect of supervised exercise on hyper-kyphosis using the Debrunner Kyphometer, a non-radiologic gold standard tool. This device measures the kyphosis angle by positioning its arms on the spinous processes of T2-T3 (upper point) and T11-T12 (lower point), with direct angle readings from the calibrated scale. Measurements are taken in degrees, with hyper-kyphosis defined as ≥53° in women and ≥55° in men.
Rate of changes in forward head posture | Pre-intervention and Week 12
  Evaluating the effect of supervised exercise on forward head posture craniocervical angle (CVA) analysis using digital photogrammetry. Reflective markers are placed on the C7 spinous process and the tragus of the ear, followed by lateral image capture at a standardized 1.5-meter distance. Image analysis software, such as Kinovea, automatically calculates the CVA angle. A normal posture is defined as CVA ≥53°, while a severe forward head posture is <50°.

SECONDARY OUTCOMES:
Change in Quality of Life (SF-36) | Pre-intervention and Week 12
  Evaluating improvements in quality of life using the Kidney Disease Quality of Life 36-item survey (KDQOL-36) questionnaire. For all KDQOL-36 subscales, scores range from 0 to 100, with higher scores consistently indicating better health-related quality of life outcomes.
Change in Fatigue Severity | Pre-intervention and Week 12
  Measuring fatigue levels before and after the intervention using Fatigue Severity Scale (FSS) (9 items on a Likert scale 1-7 (total range 9-63); Score interpretation: ≥36 indicates clinical fatigue, ≤18 indicates no fatigue. ICC = 0.91). Higher scores indicate greater fatigue.
Rate of changes of daily physical activity level | Pre-intervention and Week 12
  Assessing the effect of supervised exercise on daily activity levels using the LowPAQ questionnaire which evaluates physical activity across occupational, transportation, household, leisure, and sedentary domains, with scoring in MET-minutes per week for light (3.3 MET), moderate (4.0 MET), and vigorous (8.0 MET) activities. Activity levels are categorized as low (<600 MET-min/week), active (600-3000 MET-min/week), and highly active (>3000 MET-min/week), aligned with WHO guidelines.
Change in Muscle Strength | Pre-intervention and Week 12
  To evaluate the impact of the intervention on muscle strength using handheld dynamometry.
  Handheld dynamometry is a quantitative method for measuring isometric muscle strength. The device records maximal force exerted by the patient in standardized positions. It is portable and has shown high intra- and inter-rater reliability. The full assessment typically takes 15-20 minutes and includes major muscle groups involved in posture and mobility.
Rate of changes of balance and fall risk | Pre-intervention and Week 12
  Assessing balance improvements and fall risk reduction using Timed Up and Go (TUG) Test duration (unit: seconds, Time required to rise, walk 3 meters, turn, and return; diagnostic threshold ≥12 seconds indicates fall risk).
Rate of changes of physical function | Pre-intervention and Week 12
  Evaluating physical function improvement using the 6-minute walk test (6MWT), which measures the maximum distance covered in 6 minutes (unit: meters). Reference values: 400-700 meters for older adults and 150-346 meters for heart failure patients.
Number of participants with abnormal hematological test results | Baseline, Week 6, and Week 12
  Abnormal values will be defined based on standard lab reference ranges for Hgb, WBC, and Plt. Outcome reported as number of participants with ≥1 abnormal value.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Study Director — Pardis Specialized Wellness Institute
Locations (1):
- Pardis specialized wellness institute, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article, after deidentification are to be shared
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Not applicable. It will be accessible for public.

REFERENCES:
- [Background] Akshintala S, Khalil N, Yohay K, Muzikansky A, Allen J, Yaffe A, Gross AM, Fisher MJ, Blakeley JO, Oberlander B, Pudel M, Engelson C, Obletz J, Mitchell C, Widemann BC, Stevenson DA, Plotkin SR; REiNS International Collaboration. Reliability of Handheld Dynamometry to Measure Focal Muscle Weakness in Neurofibromatosis Types 1 and 2. Neurology. 2021 Aug 17;97(7 Suppl 1):S99-S110. doi: 10.1212/WNL.0000000000012439. Epub 2021 Jul 6. PMID 34230196
- [Background] Altintas B, Giri N, McReynolds LJ, Best A, Alter BP. Genotype-phenotype and outcome associations in patients with Fanconi anemia: the National Cancer Institute cohort. Haematologica. 2023 Jan 1;108(1):69-82. doi: 10.3324/haematol.2021.279981. PMID 35417938
- [Background] Eghbali A, Safdari SM, Yousefi Roozbahani M, Tavajohi K, Hosseini S. Fanconi Anemia: Challenges in Diagnosis and Management-A Case Series Report. Clin Case Rep. 2024 Nov 17;12(11):e9583. doi: 10.1002/ccr3.9583. eCollection 2024 Nov. PMID 39559288
- [Background] Dufour C, Pierri F. Modern management of Fanconi anemia. Hematology Am Soc Hematol Educ Program. 2022 Dec 9;2022(1):649-657. doi: 10.1182/hematology.2022000393. PMID 36485157
- [Background] Hardy SE, Gill TM. Factors associated with recovery of independence among newly disabled older persons. Arch Intern Med. 2005 Jan 10;165(1):106-12. doi: 10.1001/archinte.165.1.106. PMID 15642885
- [Background] Impellizzeri FM, Agosti F, De Col A, Sartorio A. Psychometric properties of the Fatigue Severity Scale in obese patients. Health Qual Life Outcomes. 2013 Mar 6;11:32. doi: 10.1186/1477-7525-11-32. PMID 23496886
- [Background] Moreno OM, Paredes AC, Suarez-Obando F, Rojas A. An update on Fanconi anemia: Clinical, cytogenetic and molecular approaches (Review). Biomed Rep. 2021 Sep;15(3):74. doi: 10.3892/br.2021.1450. Epub 2021 Jul 15. PMID 34405046
- [Background] Singla D, Veqar Z. Association Between Forward Head, Rounded Shoulders, and Increased Thoracic Kyphosis: A Review of the Literature. J Chiropr Med. 2017 Sep;16(3):220-229. doi: 10.1016/j.jcm.2017.03.004. Epub 2017 Sep 28. PMID 29097952
- [Background] Rayi A, Hozayen S. Chromosome Instability Syndromes. 2022 Sep 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537198/ PMID 30725883
- [Background] Wardyn GG, Rennard SI, Brusnahan SK, McGuire TR, Carlson ML, Smith LM, McGranaghan S, Sharp JG. Effects of exercise on hematological parameters, circulating side population cells, and cytokines. Exp Hematol. 2008 Feb;36(2):216-23. doi: 10.1016/j.exphem.2007.10.003. PMID 18206729
- [Background] Ye M, Liu T, Mao X, Tan X, Wang J, Xu M. Effectiveness of exercise rehabilitation on aplastic anemia patients receiving hematopoietic stem cell transplantation: study protocol for a randomized controlled trial. Trials. 2024 Jun 5;25(1):361. doi: 10.1186/s13063-024-08197-4. PMID 38840199